CLINICAL TRIAL: NCT07364266
Title: Analgesic Amputation for Algodystrophy: Feedback From a Case Series
Acronym: AMPUTALGO
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC25.0239 - AMPUTALGO
Record Dates: First submitted 2026-01-08; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Algoneurodystrophy; Amputation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- amputation for algodystrophy: A population of patients who underwent lower- or upper-limb amputation for post-traumatic algodystrophy, managed at Brest University Hospital (CHRU de Brest) between 2010 and 2025. **Inclusion criteria:**
  * Adult patients at the time of amputation;
  * Post-traumatic algodystrophy diagnosed clinically and confirmed by imaging if necessary, according to the **Budapest criteria**;
  * Amputation performed for analgesic purposes after failure of conventional medical and rehabilitation treatments;
  * Postoperative follow-up performed at **CHRU de Brest**, with available data on prosthetic fitting and postoperative activities;
  * Complete medical record accessible via the hospital electronic medical record.
  Interventions: Other: describe the time interval between amputation for post-traumatic algodystrophy and functional prosthetic fitting of the amputated limb

INTERVENTIONS:
Other: describe the time interval between amputation for post-traumatic algodystrophy and functional prosthetic fitting of the amputated limb — Primary objective endpoint: time interval, expressed in days, between the date of the amputation surgery and the date of the first effective fitting of a functional prosthesis, as documented in the medical record or during follow-up consultations.

SUMMARY:
What is the aim of the research? The study aims to describe the time interval between amputation for post-traumatic complex regional pain syndrome (CRPS) and functional prosthetic fitting of the amputated limb, within a series of patients managed in an expert center after failure of conventional treatments, in order to improve knowledge and medical practices in this field.

What data are used? The data used in this study come from your medical record. They include administrative information (age, sex, date of hospitalization, department, length of stay), medical information (diagnoses, surgical procedures, operative and consultation reports), follow-up information (functional progress, return to activities, occurrence of complications), rehabilitation and prosthetic fitting information (dates of prosthesis fitting, whether it was accepted or not, functional rehabilitation), and information from pain centers if present in the hospital medical record.

These data will be pseudonymized; that is, they will be coded and will not include your first or last name. They will be processed confidentially, only by authorized members of the research team, for exclusively scientific purposes.

Who will receive the data? Authorized members of the research team who carry out the analyses will have access to the study data in coordination with the scientific lead. All these individuals are bound by professional secrecy and confidentiality. The results of the analyses will be published in scientific journals or presented at conferences. They will always be reported in aggregate form, so that it will be completely impossible to identify a study participant.

How is the study conducted and how is your data security ensured? A computerized file containing only the data strictly necessary for the study will be created within Brest University Hospital (CHU de Brest). Your first and last names will not appear in this file.

Only authorized members of the research team will be able to access the data. Access to the database will be secured by an individual password. Analyses will always be carried out confidentially. No individual data will be extracted from the database.

The results of the study will help improve current knowledge and optimize the care of patients who may experience the same medical situation as the one you have experienced.

Your health data collected as part of this research will be kept and archived for a maximum of 5 years after the end of the study.

DETAILED DESCRIPTION:
Post-traumatic algodystrophy, or complex regional pain syndrome (CRPS) type I, is a severe and disabling complication that is often refractory to standard treatments, including rehabilitation, pharmacological therapies, and management in a pain center. In rare, extreme cases, some patients-after a long and unsuccessful therapeutic course-request amputation in order to end their chronic suffering. Although this indication remains exceptional and is overseen through multidisciplinary expert assessment, it raises major questions regarding its functional, psychological, and social benefits. To date, the literature is limited to a few isolated case reports, with no clear consensus on outcomes after amputation, particularly with respect to the time to rehabilitation and return to activities.

This retrospective study aims to describe, within a unique case series in France, the time from amputation to prosthetic fitting, as well as the time to resumption of sporting or leisure activities. Its main objective is to improve understanding of the post-amputation pathway in this atypical indication. Analysis of these data will provide points for reflection for multidisciplinary teams faced with these situations, and may potentially help guide management recommendations.

The expected benefit is:

medical: improved assessment of the benefit-risk balance of amputation in the context of CRPS scientific: addressing a gap in the literature with the largest case series published to date organizational: optimization of care pathways and reduction of delays to prosthetic fitting This study therefore fully aligns with an approach aimed at improving the quality of care for these complex patients.

This is a **retrospective observational study**, based on the analysis of existing medical data collected from a consecutive case series of patients who underwent limb amputation for post-traumatic algodystrophy, between **2010 and 2025** at **Brest University Hospital (CHRU de Brest)**. The design is **historical longitudinal**, as the data are analyzed chronologically from the amputation through postoperative follow-up, including prosthetic fitting and return to activities. **No comparison with a control group is planned**, as the objective is **descriptive**, not comparative.

This design choice is justified by the rarity of the clinical situation studied, making the construction of a control group of limited relevance, or even ethically questionable. Nevertheless, the case series makes it possible to document in detail the timeframes and post-amputation trajectories in a highly specific context that is still poorly described in the literature.

The **primary endpoint** is the time interval between the **date of amputation** and the date of **functional prosthetic fitting** (first fitting of a prosthesis). **Secondary endpoints** include the time to resumption of a physical or leisure activity, as well as the occurrence of complications (e.g., persistent pain, wound-healing problems, prosthetic fitting failures). These data are extracted from medical records and follow-up consultation reports.

No estimates of association measures (such as odds ratios or relative risks) are planned, as the study does not aim to demonstrate causality but rather to describe a care pathway and its timelines. The main advantage of this design is its feasibility in the context of a small sample size and its informative value for clinicians facing complex decisions in cases of refractory algodystrophy.

* Primary objective:** to describe the time interval between amputation for post-traumatic algodystrophy and functional prosthetic fitting of the amputated limb, within a case series of patients managed in an expert center after failure of conventional treatments.
* Primary objective endpoint:** time interval, expressed in days, between the date of the amputation surgery and the date of the first effective fitting of a functional prosthesis, as documented in the medical record or during follow-up consultations.

  * Secondary objectives

    * Assess the time interval between amputation and return to a physical or leisure activity, in order to better understand the medium-term functional impact after amputation for algodystrophy.

    * Describe the occurrence and nature of postoperative complications in these patients, including residual pain (stump pain, phantom limb pain), prosthetic fitting difficulties, and surgical complications.
    * Explore factors likely to influence time to prosthetic fitting or return to activity, such as age, sex, level of amputation, duration of algodystrophy, and prior management.
  * Measurement criteria for secondary objectives

    * Time to return to a physical or leisure activity, expressed in days from the date of amputation, as reported in consultation notes.
    * Occurrence of postoperative complications, including:
    * residual pain (stump pain, phantom limb pain),
    * prosthetic fitting difficulties or failure (non-acceptance or inability to wear the prosthesis),
    * surgical complications (delayed wound healing, infections, reoperations).
    * Analysis of factors such as age, sex, level of amputation, duration of algodystrophy, and prior management.

Description and justification of the study population

### Target population

The study concerns a population of patients who underwent **lower- or upper-limb amputation** for post-traumatic algodystrophy, managed at **CHRU de Brest** between 2010 and 2025. This rare and specific indication relies on a multidisciplinary medical decision after a prolonged pathway in a pain center, justifying rigorous and homogeneous population selection.

* Inclusion criteria

  * Adult patients at the time of amputation;

  * Post-traumatic algodystrophy diagnosed clinically and confirmed by imaging if necessary, according to the **Budapest criteria**;
  * Amputation performed for analgesic purposes, after failure of conventional medical and rehabilitation treatments;
  * Postoperative follow-up carried out at CHRU de Brest, with available data on prosthetic fitting and postoperative activities;
  * Complete medical record accessible via the hospital electronic medical record.
* Exclusion criteria

  * Patients amputated for another cause (vascular, tumor, infectious, etc.);

  * Patients not followed after amputation or immediately lost to follow-up after surgery;

  * Incomplete medical records regarding the main variables of interest (dates of amputation, prosthetic fitting, functional follow-up).
* Geographic scope

The study is **single-center**, limited to CHRU de Brest, the only facility that centralized this type of care in the region over the study period. This choice ensures homogeneity of medical practices, diagnostic criteria, and therapeutic strategy.

* Targeting and data extraction period

  * **Targeting period:** January 2010 to May 2025, corresponding to the period during which patients could be identified as having undergone an amputation for algodystrophy in the orthopedic surgery department.
  * **Data extraction period:** 2010 to June 2025, to allow analysis of the complete post-amputation pathway, including time to prosthetic fitting and return to activity, up to the most recent consultations.
* Justification of the population and collected data

The target population is small but consistent with the study objectives, which aim for an in-depth descriptive analysis of a rare yet clinically significant case series. No random sampling is planned: **all patients meeting the inclusion criteria will be included**, ensuring completeness in this low-volume context. The series is expected to include approximately **10 to 15 cases**, representing-according to the literature-one of the largest case series published to date for this indication.

Collected data will be strictly limited to variables necessary to analyze the endpoints (dates of surgery, prosthetic fitting, return to activity, complications), as well as a few targeting variables (age, sex, date of the initial trauma, amputation level) useful for exploring factors potentially associated with rehabilitation timelines. No sensitive, non-justified variables (ethnic origin, municipality of residence) will be collected. All data will be pseudonymized, with a correspondence table stored in a secure location and accessible only to authorized investigators.

This framework ensures proportionate and relevant use of personal data with respect to the scientific aims, while complying with ethical and regulatory requirements (in particular, the **GDPR**).

---

## 3.3. Population size

The study will involve a retrospective case series of patients who underwent limb amputation for analgesic purposes due to post-traumatic algodystrophy at CHRU de Brest between 2010 and 2025.

### Estimated population size

Based on an initial census conducted with the supervising team (Professor Frédéric Dubrana), approximately **10 to 15 patients** strictly meeting the inclusion criteria were managed during this period in the orthopedic surgery department. This is a realistic and exhaustive estimate in a highly specific and rare context, where amputation for algodystrophy represents a last resort after prolonged therapeutic failure.

### Epidemiological context

Post-traumatic algodystrophy (or CRPS type I) has an estimated incidence of **5 to 26 cases per 100,000 inhabitants per year**, according to international literature (de Mos et al., 2007; Bruehl, 2010). The vast majority of cases improve with conservative treatment. Chronic and severe forms are rare, and cases progressing to amputation are exceptional, generally reported as isolated case reports in the literature.

In France, there is currently no exhaustive epidemiological database specifically listing amputations for algodystrophy. Exploring national databases (ScanSanté, Open Damir) using ICD-10 codes **T79.6** (algodystrophy) or **M89.0** (algoneurodystrophic osteonecrosis) does not specifically isolate this indication for amputation. However, reports from the **HAS** and recommendations from the **SFETD** (French Society for the Study and Treatment of Pain) confirm its extreme rarity and the absence of a clear therapeutic consensus.

### Scientific justification

In this context, even a small sample of 10 to 15 patients represents a valuable source of clinical data, potentially the largest published case series to date for this indication. This number is therefore appropriate and sufficient given the purely descriptive objectives of the study (analysis of time to prosthetic fitting and return to activities), with no comparative aim or complex statistical inference. The small size is an inherent constraint linked to the nature of the condition and the therapeutic indication, and it fully justifies the choice of a retrospective observational design. Compared with the available literature (mostly case reports), our Brest series would be the largest in terms of sample size.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients at the time of amputation; Post-traumatic algodystrophy diagnosed clinically and confirmed by imaging if necessary, according to the Budapest criteria; Amputation performed for analgesic purposes, after failure of conventional medical and rehabilitation treatments; Postoperative follow-up carried out at CHRU de Brest, with available data on prosthetic fitting and postoperative activities; Complete medical record accessible via the hospital electronic medical record.

Exclusion Criteria:

* Patients amputated for another cause (vascular, tumor, infectious, etc.); Patients not followed after amputation or immediately lost to follow-up after surgery; Incomplete medical records regarding the main variables of interest (dates of amputation, prosthetic fitting, functional follow-up).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study concerns a population of patients who underwent lower- or upper-limb amputation for post-traumatic algodystrophy, managed at CHRU de Brest between 2010 and 2025. This rare and specific indication relies on a multidisciplinary medical decision after a prolonged pathway in a pain center, justifying rigorous and homogeneous population selection.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
describe the time interval between amputation for post-traumatic algodystrophy and functional prosthetic fitting of the amputated limb | 2010 to 2025
  time interval, expressed in days, between the date of the amputation surgery and the date of the first effective fitting of a functional prosthesis, as documented in the medical record or during follow-up consultations.

SECONDARY OUTCOMES:
Assess the time interval between amputation and return to a physical or leisure activity, in order to better understand the medium-term functional impact after amputation for algodystrophy. | 2010 to 2025
  Time to return to a physical or leisure activity, expressed in days from the date of amputation, as reported in consultation notes.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Chu Brest, Brest
  - CHU de Brest, Brest

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement